CLINICAL TRIAL: NCT04506645
Title: A Randomized, Double-Blind, Placebo-Controlled, Two-Part Single Ascending Dose Study to Assess the Safety, Tolerability, and Pharmacokinetics of REGN5381 (an NPR1 Agonist) in Humans
Brief Title: Study to Assess the Safety, Tolerability, and Pharmacokinetics of REGN5381 (an NPR1 Agonist) in Adult Humans
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R5381-HV-1987; 2020-000940-75 (EudraCT Number)
Record Dates: First submitted 2020-07-28; First posted 2020-08-10 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Healthy
Keywords: Normal Blood Pressure (BP); Mildly Elevated BP

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- REGN5381 (Experimental): Single dose REGN5381 administered via IV infusion
  Interventions: Drug: REGN5381
- Placebo (Other): Placebo matching single dose REGN 5381 administered via IV infusion
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: REGN5381 — Single dose REGN5381 administered via IV infusion
  Arms: REGN5381
Other: Placebo — Placebo matching single dose REGN 5381 administered via IV infusion
  Arms: Placebo

SUMMARY:
The primary objective of the study is to evaluate the safety and tolerability of single intravenous (IV) doses of REGN5381 in healthy normotensive and otherwise healthy hypertensive adults.

The secondary objectives of the study are:

* To evaluate the effect of single IV doses of REGN5381 on blood pressure (BP) and heart rate (HR) in healthy normotensive and otherwise healthy hypertensive adults
* To evaluate the effect of single IV doses of REGN5381 on cardiac stroke volume (SV)
* To evaluate the pharmacokinetics (PK) of single IV doses of REGN5381
* To evaluate the immunogenicity of single IV doses of REGN5381

ELIGIBILITY:
Inclusion Criteria:

1. Normal or mildly elevated blood pressure as defined in the protocol

Exclusion Criteria:

1. History of cardiovascular disease as defined in the protocol
2. Protocol-defined risk factors for cardiovascular disease
3. History of unexplained syncope, autonomic dysfunction, or neurologic disease.

NOTE: Additional Inclusion / Exclusion criteria apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-12-14 (Actual); Study Completion 2022-12-14 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Up to Day 78

SECONDARY OUTCOMES:
Change from baseline in Systolic Blood Pressure (SBP) | Up to Day 78
Change from baseline in Diastolic Blood Pressure (DBP) | Up to Day 78
Change from baseline in Mean Arterial Pressure (MAP) | Baseline to Day 4
Change from baseline in Pulse Pressure (PP) | Baseline to Day 4
Change from baseline in Heart Rate (HR) | Up to Day 78
Change from baseline in Stroke Volume (SV) | Baseline to Day 4
Maximum change from baseline in SBP across the first 24 hours postdose | Baseline to Day 2 (24-hours post dose)
Maximum change from baseline in DBP across the first 24 hours postdose | Baseline to Day 2 (24-hours post dose)
Maximum change from baseline in MAP across the first 24 hours postdose | Baseline to Day 2 (24-hours post dose)
Maximum change from baseline in PP across the first 24 hours postdose | Baseline to Day 2 (24-hours post dose)
Maximum change from baseline in HR across the first 24 hours postdose | Baseline to Day 2 (24-hours post dose)
Maximum change from baseline in SV across the first 24 hours postdose | Baseline to Day 2 (24-hours post dose)
Change from baseline in the 24-hour mean SBP measured from 0 to 24 hours, 24 to 48 hours, and 48 to 72 hours postdose | Baseline to 24 hours postdose, 24 hours to 48 hours postdose, 48 hours to 72 hours postdose
  Baseline 24-hour mean SBP is measured from 0 to 24 hours pre-dose
Change from baseline in the 24-hour mean DBP measured from 0 to 24 hours, 24 to 48 hours, and 48 to 72 hours postdose | Baseline to 24 hours, 24 to 48 hours, and 48 to 72 hours postdose
  Baseline 24-hour mean DBP is measured from 0 to 24 hours pre-dose
Change from baseline in the 24-hour mean MAP measured from 0 to 24 hours, 24 to 48 hours, and 48 to 72 hours postdose | Baseline to 24 hours, 24 to 48 hours, and 48 to 72 hours postdose
  Baseline 24-hour mean MAP is measured from 0 to 24 hours pre-dose
Change from baseline in the 24-hour mean PP measured from 0 to 24 hours, 24 to 48 hours, and 48 to 72 hours postdose | Baseline to 24 hours, 24 to 48 hours, and 48 to 72 hours postdose
  Baseline 24-hour mean PP is measured from 0 to 24 hours pre-dose
Change from baseline in the 24-hour mean HR measured from 0 to 24 hours, 24 to 48 hours, and 48 to 72 hours postdose | Baseline to 24 hours, 24 to 48 hours, and 48 to 72 hours postdose
  Baseline 24-hour mean HR is measured from 0 to 24 hours pre-dose
Concentrations of REGN5381 over time | Up to Day 78
Number of subjects who develop anti-drug antibodies (ADA) and titers | Up to Day 78
Percentage of subjects who develop anti-drug antibodies (ADA) and titers | Up to Day 78

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (2):
- Belgium (2):
  - Ghent University, Ghent
  - Universitair Ziekenhuis Leuven Gasthuisberg Campus, Leuven

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Individual anonymized participant data will be considered for sharing once the indication has been approved by a regulatory body, if there is legal authority to share the data and there is not a reasonable likelihood of participant re-identification.
Access Criteria: Qualified researchers may request access to anonymized patient level data or aggregate study data when Regeneron has received marketing authorization from major health authorities (e.g., Food and Drug Administration (FDA), European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc) for the product and indication, has the legal authority to share the data, and has made the study results publicly available (eg, scientific publication, scientific conference, clinical trial registry).
URL: https://vivli.org/